CLINICAL TRIAL: NCT03925142
Title: Effects of Replacing Starchy Vegetables and Refined Grains With Beef in a Vegetarian Diet on Cardio-metabolic Disease Risk Factors
Brief Title: Effects of Replacing Starchy Vegetables and Refined Grains With Beef on Cardio-metabolic Disease Risk Factors (S53)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Wayne Campbell, Principal Investigator, Purdue University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 1809021091
Record Dates: First submitted 2019-04-09; First posted 2019-04-24 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-12

CONDITIONS: Diet Modification
Keywords: beef; cardio-metabolic disease

STUDY DESIGN:
Intervention Model Description: This is a 16-week randomized, cross-over, controlled, single-blind study. During weeks 1 and 11, participant's usual, unrestricted dietary intakes will be assessed. At week 2, they will be randomized and assigned to consume either the controlled lacto-ovo vegetarian diet or beef diet for the first 5-week dietary intervention during weeks 2-6. They will consume the other diet during weeks 12-16. Two fasting-state serum samples and one stool samples will be collected during study weeks 1,6,11, and 16.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Controlled healthy vegetarian diet (Active Comparator): Subjects will be randomized and assigned to consume the controlled Healthy Vegetarian Eeating Pattern for 5 weeks.
  Interventions: Other: Controlled healthy vegetarian diet
- Controlled beef diet (Experimental): Subjects will be randomized and assigned to consume the beef diet for 5 weeks, which will substitute predominantly starchy vegetables and refined grains with 6 oz. of lean unprocessed beef/day.
  Interventions: Other: Controlled beef diet

INTERVENTIONS:
Other: Controlled healthy vegetarian diet — The controlled healthy vegetarian diet will follow the Dietary Guidelines for American's recommendations. All foods and beverages will be provided during intervention to achieve the desired eating pattern.
  Arms: Controlled healthy vegetarian diet
Other: Controlled beef diet — The controlled beef diet will incorporate various cuts of lean unprocessed red meat into the healthy vegetarian eating pattern, as approved by the American Heart Association's Food Certification Program. The beef diet will isocalorically replace starchy vegetables and/or refined grains with 6 oz. of beef/day for five weeks.
  Arms: Controlled beef diet

SUMMARY:
The purpose of this study is to assess the effects of replacing starchy vegetables and refined grains with beef in a vegetarian diet on cardio-metabolic disease risk factors in adults in a cross-over, randomized controlled feeding trial.

DETAILED DESCRIPTION:
The purpose of this study is to assess the effects of replacing starchy vegetables and refined grains with beef in a vegetarian diet on cardio-metabolic disease risk factors in adults in a cross-over, randomized controlled feeding trial. The hypothesis is that isocalorically replacing predominantly starchy vegetables and refined grains with 6 oz. of beef/day will enhance improvements in cardiometabolic disease risk factors, particularly atherosclerotic-promoting lipids and lipoproteins. It is also hypothesized that participant satisfaction and acceptance of a healthy eating pattern with 6 oz. of beef per day will be higher compared to without beef.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* 30-69 years old
* BMI 25-37 kg/m2
* Total cholesterol <260 mg/dL
* Low-density lipoprotein cholesterol <190 mg/dL
* Glucose <110 mg/dL
* Systolic/diastolic blood pressure < 140/90
* Body weight stable for 3 months prior (±3 kg)
* Stable physical activity regimen 3 months prior
* Medication use stable for 6 months prior
* Non-smoking
* Not drinking more than 2 alcoholic drinks per day
* Non-diabetic
* Not lactose-intolerant
* Not acutely ill
* Non-pregnant and not lactating.
* Participants must be willing and able to consume the prescribed diets (lacto-ovo vegetarian and omnivorous).

Exclusion Criteria:

* <30 or >69 years old
* BMI <25.0 or >37 kg/m2
* Fasting serum total cholesterol > 260 mg/dL
* Low-density lipoprotein cholesterol >189 mg/dL
* Glucose >110 mg/dL
* Systolic/diastolic blood pressure > 140/90
* Body weight stable for <3 months prior (±3 kg)
* Stable physical activity regimen < 3 months prior
* Medication use unstable for 6 months prior and using medications
* Smoking
* Drinking more than 2 alcoholic drinks per day
* Diabetic
* Have renal failure
* Have liver failure
* Have cardiovascular events (myocardial infarction or stroke) during the 6 months prior to the study
* Pregnant or lactating

Ages: 30 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2019-06-04 (Actual); Primary Completion 2021-10-28 (Actual); Study Completion 2021-10-28 (Actual)

PRIMARY OUTCOMES:
Concentrations of serum lipids, lipoproteins, and total apolipoprotein B | 1.5 years
  The hypothesis is that substituting starchy vegetables and refined grain with lean unprocessed beef in a plant based eating pattern will result in greater reduction in the concentrations of low-density lipoprotein-cholesterol, total cholesterol, triglycerides, and total apolipoprotein B, but greater increase in concentration of high-density lipoprotein-cholesterol.

SECONDARY OUTCOMES:
Level of fasting blood pressure | 1.5 years
  The hypothesis is that substituting starchy vegetables and refined grain with lean unprocessed beef in a plantbased eating pattern will result in greater reductions in fasting blood pressure.
Level of fasting serum insulin | 1.5 years
  The hypothesis is that substituting starchy vegetables and refined grain with lean unprocessed beef in a plantbased eating pattern will result in greater reductions in fasting serum insulin.
Concentration of fasting serum glucose | 1.5 years
  The hypothesis is that substituting starchy vegetables and refined grain with lean unprocessed beef in a plantbased eating pattern will result in greater reductions in fasting serum glucose.
Size of lipoprotein particle | 1.5 years
  The hypothesis is that substituting starchy vegetables and refined grain with lean unprocessed beef in a plantbased eating pattern will result in greater reductions in low-density lipoprotein particle size.

OTHER OUTCOMES:
Questionnaire score of consumer satisfaction of a plant-based eating pattern | 1.5 years
  The hypothesis is that substituting starchy vegetables and refined grain with lean unprocessed beef in a plant-based eating pattern will result in a higher score of consumer satisfaction using the Dietary Satisfaction Questionnaire designed by study investigators. The Dietary Satisfaction Questionnaire is a six-point Likert scale ranging from "strongly disagree" to "strongly agree". The questionnaire includes 23 questions on overall satisfaction of different aspects of the intervention diets, such as fullness after meals, enjoyment of study foods, and impact of study foods on personal well-being. The Likert scale will be matched to numerical values for scoring (0=strongly disagree, 1=disagree, 2=slightly disagree, 3=slightly agree, 4=agree, 5=strongly agree). Total score ranges from 0 to 115 and higher score represents higher dietary satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Wayne W Campbell, PhD, Principal Investigator — Purdue University
Locations (1):
- Purdue University, West Lafayette, Indiana, United States